CLINICAL TRIAL: NCT02315352
Title: Randomized, Single Blind, Cross-over Study to Evaluate the Palatability of New Orally Disintegrating Tablets of PZQ and L-PZQ Versus Current PZQ Tablets in African Children Age 6-11 Years
Brief Title: Cross-over Study to Evaluate the Palatability of New Orally Disintegrating Tablets (ODTs) of Praziquantel (PZQ) and L-PZQ Versus Current PZQ Tablets in African Children Age 6-11 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EMR200661-002
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Healthy; L-PZQ; PZQ; MSC2499550A; Praziquantel
MeSH Terms: interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 and 2 (Experimental): A-B or B-A where A: L-PZQ ODT (MSC 2499550A) put on tongue; B: Rac-PZQ ODT (MSC1028703A) put on the tongue
  Interventions: Drug: L-PZQ ODT; Drug: Rac-PZQ ODT
- Period 3, 4 and 5 (Experimental): C-D-E; C-E-D; D-E-C; D-C-E; E-C-D; E-D-C where C: L-PZQ ODT (MSC 2499550A) dispersed in water; D: Rac-PZQ ODT (MSC1028703A) dispersed in water; E: Cesol® 150 mg crushed in water
  Interventions: Drug: L-PZQ ODT; Drug: Rac-PZQ ODT; Drug: Cesol®

INTERVENTIONS:
Drug: L-PZQ ODT — L-PZQ ODT (MSC2499550A) tablet at a dose of 150 milligram (mg) put and disintegrated in the mouth without water
  Other Names: MSC 2499550A
  Arms: Period 1 and 2
Drug: Rac-PZQ ODT — Rac-PZQ ODT (MSC1028703A) tablet at a dose of 150 mg put and disintegrated in the mouth without water
  Other Names: MSC1028703
  Arms: Period 1 and 2
Drug: L-PZQ ODT — L-PZQ (MSC2499550A) tablet at a dose of 150 mg dispersed in water
  Other Names: MSC 2499550A
  Arms: Period 3, 4 and 5
Drug: Rac-PZQ ODT — Rac-PZQ ODT (MSC1028703A) tablet at a dose of 150 mg dispersed in water
  Other Names: MSC1028703A
  Arms: Period 3, 4 and 5
Drug: Cesol® — Cesol® tablet at a dose of 150 mg crushed in water
  Other Names: PZQ
  Arms: Period 3, 4 and 5

SUMMARY:
The primary objective of the trial is to compare the "overall palatability" of the new orally disintegrating L-Praziquantel (L-PZQ ODT), the new racemate PZQ ODT (Rac-PZQ ODT) and the current available racemate PZQ tablets (reference) as assessed by means of human gustatory sensation tests (100 millimeter [mm] visual analogue scale [VAS] scoring modified by the incorporation of a 5 point facial hedonic scale).

The secondary objectives are

* To obtain feedback from children regarding the taste of different formulations using an open ended questionnaire
* To document any discomfort or other observation in relation to acceptance of the study medication

DETAILED DESCRIPTION:
Initially pupils will be invited with their parents to school where they will be asked to give consent/assent in to the study and they will be instructed on how to follow up the taste study procedures. Enrollments will occur in the health facilities in Ikwiriri/Kibiti at the end of successive training. Informed consent from parents and guardians and assent from the child will be obtained before participation in the study. The study will be conducted in school children 6 years and older as recommended by the Committee for medical product for human use (CHMP) reflection paper: formulations of choice for the pediatric population.

-This is a randomized, five-period cross over, single center swill and spit taste study where the drug will not be swallowed but will be spit out after tasting.

On Day 1, the subjects will assess the palatability of the following arms in a randomized sequence:

* L-PZQ ODT (150 mg) put and disintegrated in the mouth
* Rac- PZQ ODT (150 mg) put and disintegrated in the mouth

On Day 2, the subjects will assess the palatability of the following arms in a randomized sequence:

* L-PZQ ODT (150 mg) dispersed in water administered in the mouth cavity
* Rac- ODT (150 mg) dispersed in water administered in the mouth cavity
* 150 mg current PZQ tablet (1/4 of a 600 mg tablet) crushed, dispersed in water and administered in the mouth cavity

Gustatory sensation studies will be performed on the different formulations immediately after tasting and 2-5 min after the study drug has been spat out.

All volunteers will be asked to place a mark along the line with the use of a 100 mm visual analogue scale (VAS) that incorporates a 5 points hedonic scale for "overall palatability".

In addition, any discomfort or other observation in relation to acceptance of the study medication (Example: spitting out of the medicine) will be reported by the parents or investigator.

An open ended questionnaire (description of mouth feeling and taste description) will be conducted for each child during the washout period. After the trial a therapeutic dose of Praziquantel will be made available to the local health council and management team to provide to the participating school.

ELIGIBILITY:
Inclusion criteria:

1. Children male or female aged 6-11 years (inclusive)
2. Parents or guardians gave written informed consent prior to any trial related procedure and child gave assent
3. Able to communicate well with the Investigator, understanding the protocol requirements and restrictions, and willing to comply with the requirements of the entire trial
4. Subjects should be able to hold 2 milliliter (mL) of any appropriate juice in their mouth for 10 seconds without swallowing it and to keep a candy in the mouth for 20 seconds without swallowing it
5. Children who are able to properly assess and differentiate flavours of different soft drinks
6. Children who are able to use a hedonic scale (children were trained before the study)

Exclusion criteria:

1. Unlikely to comply with the protocol requirements, instructions and trial-related restrictions, example: uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial
2. Children with any condition or dietary habit known to interfere with the sense of smell and taste, ingestion of any medication (except paracetamol)
3. Children with significant illness in the previous 2 weeks
4. Any surgical or medical condition, or any significant disease that in the opinion of the investigator, constitutes a risk or a contraindication for the participation of the subject in the study that could interfere with the study objectives, conduct or evaluation
5. Children who have participated in any clinical investigation within the previous 4 weeks

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Ifakara Health Institute, Ikwiriri, Rufiji, Tanzania

REFERENCES:
- [Background] CHMP. (2005). Reflection paper: formulation of choice for the paediatric population. EMA
- [Derived] Mahende MK, Huber E, Kourany-Lefoll E, Ali A, Hayward B, Bezuidenhout D, Bagchus W, Kabanywanyi AM. Comparative palatability of orally disintegrating tablets (ODTs) of Praziquantel (L-PZQ and Rac-PZQ) versus current PZQ tablet in African children: A randomized, single-blind, crossover study. PLoS Negl Trop Dis. 2021 Jun 9;15(6):e0007370. doi: 10.1371/journal.pntd.0007370. eCollection 2021 Jun. PMID 34106922

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a swill and spit taste study where the drug was not swallowed but spit out after tasting. Gustatory sensation tests were performed on the different formulations immediately after tasting and 2-5 min after the study drug has been spat out.
Groups:
- L-PZQ Then Rac-PZQ (Day 1): Subjects were administered L- Praziquantel (L-PZQ) 150 milligram (mg) oral disintegrating tablet (ODT) in first intervention period followed by racemate praziquantel (Rac-PZQ) 150 mg ODT in the second intervention period. A washout period of 1 hour was maintained between the intervention periods. The intervention was directly placed on the tongue of the subjects (without water) and the subjects were asked to spit out the tablet in a waste container. A mouth check was performed after the assessment to ensure that no particles remain in the oral cavity.
- Rac-PZQ Then L-PZQ (Day 1): Subjects were administered Rac-PZQ 150 mg ODT in first intervention period followed by L-PZQ 150 mg ODT in the second intervention period. A washout period of 1 hour was maintained between the intervention periods. The intervention was directly placed on the tongue of the subjects (without water) and the subjects were asked to spit out the tablet in a waste container. A mouth check was performed after the assessment to ensure that no particles remain in the oral cavity.
- L-PZQ Then Rac-PZQ Then Cesol® (Day 2): Subjects who were randomized to either 'L-PZQ Then Rac-PZQ' or 'Rac-PZQ Then L-PZQ' sequence on Day 1 received L-PZQ 150 mg ODT as a solution via a syringe in the buccal cavity in third intervention period followed by Rac-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in fourth intervention period and then Cesol® (currently available praziquantel tablet) 150 mg administered as a suspension via a syringe in the buccal cavity in the fifth intervention period. A washout period of 1 hour was maintained between the intervention periods. The interventions were dispersed in water and administered in the buccal cavity using a syringe. Subject was asked to hold the solution/suspension for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
- L-PZQ Then Cesol® Then Rac-PZQ (Day 2): Subjects who were randomized to either 'L-PZQ Then Rac-PZQ' or 'Rac-PZQ Then L-PZQ' sequence on Day 1 received L-PZQ 150 mg ODT as a solution via a syringe in the buccal cavity in third intervention period followed by Cesol® 150 mg administered as a suspension via a syringe in the buccal cavity in fourth intervention period and then Rac-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in the fifth intervention period. A washout period of 1 hour was maintained between the intervention periods. The interventions were dispersed in water and administered in the buccal cavity using a syringe. Subject was asked to hold the solution/suspension for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
- Rac-PZQ Then Cesol® Then L-PZQ (Day 2): Subjects who were randomized to either 'L-PZQ Then Rac-PZQ' or 'Rac-PZQ Then L-PZQ' sequence on Day 1 received Rac-PZQ 150 mg ODT as a solution via a syringe in the buccal cavity in third intervention period followed by Cesol® 150 mg administered as a suspension via a syringe in the buccal cavity in fourth intervention period and then L-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in the fifth intervention period. A washout period of 1 hour was maintained between the intervention periods. The interventions were dispersed in water and administered in the buccal cavity using a syringe. Subject was asked to hold the solution/suspension for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
- Rac-PZQ Then L-PZQ Then Cesol® (Day 2): Subjects who were randomized to either 'L-PZQ Then Rac-PZQ' or 'Rac-PZQ Then L-PZQ' sequence on Day 1 received Rac-PZQ 150 mg ODT as a solution via a syringe in the buccal cavity in third intervention period followed by L-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in fourth intervention period and then Cesol® 150 mg administered as a suspension via a syringe in the buccal cavity in the fifth intervention period. A washout period of 1 hour was maintained between the intervention periods. The interventions were dispersed in water and administered in the buccal cavity using a syringe. Subject was asked to hold the solution/suspension for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
- Cesol® Then L-PZQ Then Rac-PZQ (Day 2): Subjects who were randomized to either 'L-PZQ Then Rac-PZQ' or 'Rac-PZQ Then L-PZQ' sequence on Day 1 received Cesol® 150 mg as a suspension via a syringe in the buccal cavity in third intervention period followed by L-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in fourth intervention period and then Rac -PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in the fifth intervention period. A washout period of 1 hour was maintained between the intervention periods. The interventions were dispersed in water and administered in the buccal cavity using a syringe. Subject was asked to hold the solution/suspension for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
- Cesol® Then Rac-PZQ Then L-PZQ (Day 2): Subjects who were randomized to either 'L-PZQ Then Rac-PZQ' or 'Rac-PZQ Then L-PZQ' sequence on Day 1 received Cesol® 150 mg as a suspension via a syringe in the buccal cavity in third intervention period followed by Rac-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in fourth intervention period and then L-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in the fifth intervention period. A washout period of 1 hour was maintained between the intervention periods. The interventions were dispersed in water and administered in the buccal cavity using a syringe. Subject was asked to hold the solution/suspension for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
Period: First Intervention (Day 1)
Arm/Group | L-PZQ Then Rac-PZQ (Day 1) | Rac-PZQ Then L-PZQ (Day 1) | L-PZQ Then Rac-PZQ Then Cesol® (Day 2) | L-PZQ Then Cesol® Then Rac-PZQ (Day 2) | Rac-PZQ Then Cesol® Then L-PZQ (Day 2) | Rac-PZQ Then L-PZQ Then Cesol® (Day 2) | Cesol® Then L-PZQ Then Rac-PZQ (Day 2) | Cesol® Then Rac-PZQ Then L-PZQ (Day 2)
Started | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (Day 1)
Arm/Group | L-PZQ Then Rac-PZQ (Day 1) | Rac-PZQ Then L-PZQ (Day 1) | L-PZQ Then Rac-PZQ Then Cesol® (Day 2) | L-PZQ Then Cesol® Then Rac-PZQ (Day 2) | Rac-PZQ Then Cesol® Then L-PZQ (Day 2) | Rac-PZQ Then L-PZQ Then Cesol® (Day 2) | Cesol® Then L-PZQ Then Rac-PZQ (Day 2) | Cesol® Then Rac-PZQ Then L-PZQ (Day 2)
Started | 24 | 24 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 24 (Out of 24 subjects completing this period, 1 discontinued before assignment to any sequence on Day 2) | 24 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (Day 2)
Arm/Group | L-PZQ Then Rac-PZQ (Day 1) | Rac-PZQ Then L-PZQ (Day 1) | L-PZQ Then Rac-PZQ Then Cesol® (Day 2) | L-PZQ Then Cesol® Then Rac-PZQ (Day 2) | Rac-PZQ Then Cesol® Then L-PZQ (Day 2) | Rac-PZQ Then L-PZQ Then Cesol® (Day 2) | Cesol® Then L-PZQ Then Rac-PZQ (Day 2) | Cesol® Then Rac-PZQ Then L-PZQ (Day 2)
Started | 0 | 0 | 7 | 8 | 8 | 7 | 9 | 8
Completed | 0 | 0 | 7 | 8 | 8 | 7 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention (Day 2)
Arm/Group | L-PZQ Then Rac-PZQ (Day 1) | Rac-PZQ Then L-PZQ (Day 1) | L-PZQ Then Rac-PZQ Then Cesol® (Day 2) | L-PZQ Then Cesol® Then Rac-PZQ (Day 2) | Rac-PZQ Then Cesol® Then L-PZQ (Day 2) | Rac-PZQ Then L-PZQ Then Cesol® (Day 2) | Cesol® Then L-PZQ Then Rac-PZQ (Day 2) | Cesol® Then Rac-PZQ Then L-PZQ (Day 2)
Started | 0 | 0 | 7 | 8 | 8 | 7 | 9 | 8
Completed | 0 | 0 | 7 | 8 | 8 | 7 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Intervention (Day 2)
Arm/Group | L-PZQ Then Rac-PZQ (Day 1) | Rac-PZQ Then L-PZQ (Day 1) | L-PZQ Then Rac-PZQ Then Cesol® (Day 2) | L-PZQ Then Cesol® Then Rac-PZQ (Day 2) | Rac-PZQ Then Cesol® Then L-PZQ (Day 2) | Rac-PZQ Then L-PZQ Then Cesol® (Day 2) | Cesol® Then L-PZQ Then Rac-PZQ (Day 2) | Cesol® Then Rac-PZQ Then L-PZQ (Day 2)
Started | 0 | 0 | 7 | 8 | 8 | 7 | 9 | 8
Completed | 0 | 0 | 7 | 8 | 8 | 7 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- L-PZQ Then Rac-PZQ (Day 1): L- Praziquantel (L-PZQ) 150 milligram (mg) oral disintegrating tablet (ODT) in first intervention period followed by racemate praziquantel (Rac-PZQ) 150 mg ODT in the second intervention period. A washout period of 1 hour was maintained between the intervention periods. The intervention was directly placed on the tongue of the subjects (without water) and the subjects were asked to spit out the tablet in a waste container. A mouth check was performed after the assessment to ensure that no particles remain in the oral cavity.
- Rac-PZQ Then L-PZQ (Day 1): Rac-PZQ 150 mg ODT in first intervention period followed by L-PZQ 150 mg ODT in the second intervention period. A washout period of 1 hour was maintained between the intervention periods. The intervention was directly placed on the tongue of the subjects (without water) and the subjects were asked to spit out the tablet in a waste container. A mouth check was performed after the assessment to ensure that no particles remain in the oral cavity.
- Total: Total of all reporting groups
Arm/Group | L-PZQ Then Rac-PZQ (Day 1) | Rac-PZQ Then L-PZQ (Day 1) | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 24 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Palatability Visual Analogue Scale (VAS) Score at 0 Minute (Right After the Spit-out of the Investigational Medicinal Product [IMP])
Description: Overall palatability was assessed on a 0 to 100 unit VAS scale, where higher scores indicate better palatability.
Time Frame: 0 minute (Right After the Spit-out of the IMP)
Population: The Safety Set (SAF) included all enrolled subjects who received at least 1 dose of any study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- L-PZQ (Without Water) Day 1: All subjects who received L-PZQ 150 mg ODT directly placed on the tongue of the subjects (without water) and the subjects were asked to spit out the tablet in a waste container in any intervention period. A mouth check was performed after the assessment to ensure that no particles remain in the oral cavity.
- Rac-PZQ (Without Water) Day 1: All subjects who received Rac-PZQ 150 mg ODT directly placed on the tongue of the subjects (without water) and the subjects were asked to spit out the tablet in a waste container in any intervention period. A mouth check was performed after the assessment to ensure that no particles remain in the oral cavity.
- L-PZQ (With Water) Day 2: All subjects who received L-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in any intervention period. Subject was asked to hold the solution for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
- Rac-PZQ (With Water) Day 2: All subjects who received Rac-PZQ 150 mg ODT administered as a solution via a syringe in the buccal cavity in any intervention period. Subject was asked to hold the solution for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles remain in the oral cavity.
- Cesol® (With Water) Day 2: All subjects who received Cesol® administered as a solution via a syringe in the buccal cavity in any intervention period. Subject was asked to hold the solution for 10 sec in mouth and then spat out the liquid in a waste container. A mouth check should be performed after the administration to ensure that no particles.
Arm/Group | L-PZQ (Without Water) Day 1 | Rac-PZQ (Without Water) Day 1 | L-PZQ (With Water) Day 2 | Rac-PZQ (With Water) Day 2 | Cesol® (With Water) Day 2
Number analyzed (Participants) | 48 | 48 | 47 | 47 | 47
units on a scale | 49.0 (33.65) | 39.3 (28.43) | 67.5 (31.14) | 51.4 (32.35) | 20.3 (24.91)

2. Secondary Outcome: Overall Palatability VAS Score at 2-5 Minutes
Description: Overall palatability was assessed on a 0 to 100 unit VAS scale, where higher scores indicate better palatability.
Time Frame: 2-5 minutes (After the IMP has been spat out)
Population: The Safety Set (SAF) included all enrolled subjects who received at least 1 dose of any study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-PZQ (Without Water) Day 1 | Rac-PZQ (Without Water) Day 1 | L-PZQ (With Water) Day 2 | Rac-PZQ (With Water) Day 2 | Cesol® (With Water) Day 2
Number analyzed (Participants) | 48 | 48 | 47 | 47 | 47
units on a scale | 50.7 (27.23) | 45.1 (29.62) | 61.1 (21.19) | 50.2 (25.92) | 33.5 (22.23)

3. Secondary Outcome: Number of Subjects With Mouth Feeling and Taste Description Evaluation
Description: Mouth feeling was described in terms of "sweet", "bitter", "sticky" or "smooth" as per the experience of the subject with the trial medication.
Time Frame: 2-5 minutes (After the IMP has been spat out)
Population: The data for this outcome measure could not be evaluated as data were not collected according to protocol.
Arm/Group | L-PZQ (Without Water) Day 1 | Rac-PZQ (Without Water) Day 1 | L-PZQ (With Water) Day 2 | Rac-PZQ (With Water) Day 2 | Cesol® (With Water) Day 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Subjects With Discomfort or Observations Relating to Acceptance of the Study Medication
Time Frame: 2-5 minutes
Population: The Safety Set (SAF) included all enrolled subjects who received at least 1 dose of any study drug.
Measure: Number; unit: Subjects
Arm/Group | L-PZQ (Without Water) Day 1 | Rac-PZQ (Without Water) Day 1 | L-PZQ (With Water) Day 2 | Rac-PZQ (With Water) Day 2 | Cesol® (With Water) Day 2
Number analyzed (Participants) | 48 | 48 | 47 | 47 | 47
Subjects | 0 | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Arm/Group | L-PZQ (Without Water) Day 1 | Rac-PZQ (Without Water) Day 1 | L-PZQ (With Water) Day 2 | Rac-PZQ (With Water) Day 2 | Cesol® (With Water) Day 2
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/48 | 1/48 | 0/47 | 0/47 | 0/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-PZQ (Without Water) Day 1 (N=48) | Rac-PZQ (Without Water) Day 1 (N=48) | L-PZQ (With Water) Day 2 (N=47) | Rac-PZQ (With Water) Day 2 (N=47) | Cesol® (With Water) Day 2 (N=47)
Malaria (Infections and infestations) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No